CLINICAL TRIAL: NCT05256771
Title: Safety and Efficacy of Electrical Muscle Stimulation Combined with 1064 Nm Diode Laser, Pulsed Electromagnetic Field (PEMF) and Vacuum Assisted Radio Frequency (RF) for Non-invasive Body Contouring and Fat Reduction.
Brief Title: Electrical Muscle Stimulation with 1064 Nm Diode Laser and RF/PEMF for Non-invasive Body Contouring and Fat Reduction.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BL0221
Record Dates: First submitted 2022-02-03; First posted 2022-02-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Fat Reduction; Muscle Tone Increased
MeSH Terms: conditions — Muscle Hypertonia | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: 3 Arms at a ratio of 2:1:1 (A:B:C): Arm A: Full Treatment Arm (Laser + EMS + RF/PEMF) Arm B: EMS/RF Arm (EMS + RF/PEMF) Arm C: EMS Arm (EMS only)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded, independent photo review comparing the pre-treatment and post-treatment Follow-up 2 photographs by a physician board-certified in dermatology to evaluate contour improvement per the Global Aesthetic Improvement Scale (GAIS).
  Blinded Investigator review comparing the pre-treatment photographs and post-treatment Follow-up 1 & 2 live assessment by the Primary Investigator to evaluate contour improvement per the Global Aesthetic Improvement Scale (PI-GAIS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Arm A: Full Treatment Arm (Laser + EMS + RF/PEMF) (Active Comparator): Arm A: Three (3) diode laser treatments treatments at days 0, 28 and 56 (±2 days). Subjects will also receive bi-weekly electrical muscle stimulation and pulsed electromagnetic fields/vacuum assisted radio frequency treatments at days 0, 14, 28, 42 and 56 (±2 days).
  Interventions: Device: EMS; Device: 1064 nm diode laser; Device: RF/PEMF
- Arm B: EMS/RF Arm (EMS + RF/PEMF) (Active Comparator): Arm B: Subjects will receive bi-weekly electrical muscle stimulation and pulsed electromagnetic fields/vacuum assisted radio frequency treatments at days 0, 14, 28, 42 and 56 (±2 days).
  Interventions: Device: EMS; Device: RF/PEMF
- Arm C: EMS Arm (EMS only) (Active Comparator): Arm C: Subjects will receive weekly electrical muscle stimulation treatments at days 0, 7, 14, 21, 28 and 35 (±2 days).
  Interventions: Device: EMS

INTERVENTIONS:
Device: EMS — Abdominal muscle stimulation using EMS
Device: 1064 nm diode laser — Adipose tissue heating using 1064 nm diode laser
  Arms: Arm A: Full Treatment Arm (Laser + EMS + RF/PEMF)
Device: RF/PEMF — Collagen re-modelling and reduction in subcutaneous fat using RF/PEMF
  Arms: Arm A: Full Treatment Arm (Laser + EMS + RF/PEMF); Arm B: EMS/RF Arm (EMS + RF/PEMF)

SUMMARY:
Multi-center, three-arm, randomized, evaluator-blinded study of electrical muscle stimulation (EMS) and/or 1064 nm diode laser, pulsed electromagnetic field (PEMF) and vacuum assisted radio frequency (RF) using the Venus Bliss Max for fat reduction, body contouring and aesthetic improvement.

DETAILED DESCRIPTION:
The study will enroll up to 60 male and female subjects, ≥ 18 years of age, requesting non-invasive electrical muscle stimulation (EMS) and/or lipolysis of the abdomen and flanks. Subjects will be randomized to one of three arms as per randomization scheme.

This study will have 3 Arms at a ratio of 2:1:1 (A:B:C):

Arm A: Full Treatment Arm (Laser + EMS + RF/PEMF) Arm B: EMS/RF Arm (EMS + RF/PEMF) Arm C: EMS Arm (EMS only)

Arm A: Three (3) diode laser treatments treatments at days 0, 28 and 56 (±2 days). Subjects will also receive bi-weekly electrical muscle stimulation and pulsed electromagnetic fields (PEMF)/vacuum assisted radio frequency (RF) treatments at days 0, 14, 28, 42 and 56 (±2 days).

Arm B: Subjects will receive bi-weekly electrical muscle stimulation and pulsed electromagnetic fields/vacuum assisted radio frequency treatments at days 0, 14, 28, 42 and 56 (±2 days).

Arm C: Subjects will receive weekly electrical muscle stimulation treatments at days 0, 7, 14, 21, 28 and 35 (±2 days).

Subjects in Arms A and B will be followed at 84 and 140 days (±7 days) after their last treatment. Subjects in Arm C will be followed at 63 and 119 days (±7 days) after their last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects > 18 years of age and ≤65 years of age.
2. Subject agrees to refrain from any new abdominal training exercises during the course of the study.
3. BMI ≤ 30 kg/m2 as determined at screening.
4. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in the last 6 months, including presence of post-partum diastasis.
2. Any previous liposuction/lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months.
3. History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection) or use of immunosuppressive medications last 6 months prior to and during the course of the study.
4. History of hyperlipidemia, diabetes mellitus, hepatitis, blood coagulopathy or excessive bleeding.
5. Use of antiplatelet medications (81 mg acetylsalicylic acid daily permitted), anticoagulants, thrombolytics or anti-inflammatory medications within 2 weeks of treatment or a history of bleeding disorders.
6. History of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
7. Having a permanent implant in the treatment area such as metal plates or an injected chemical substance such as silicone or parenteral gold therapy (gold sodium thiomalate), or drug delivery system that would prevent treatment at the treatment site.
8. Use of medications, herbs, food supplements, and vitamins known to induce photosensitivity to light exposure at the wavelength used or history of photosensitivity disorder.
9. Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections.
10. Tattoos in the treatment area
11. Numbness, tingling or other altered sensation in the treatment area.
12. Known sensitivity or allergy to isopropyl alcohol and propylene glycol, hydrogel or latex or any substance used during treatments by the clinic (if applicable).
13. Unable or unwilling to comply with the study requirements.
14. Enrolled in a clinical study of any other investigational drug or device.
15. Any other condition or laboratory value that would, in the professional opinion of the Investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Blinded, independent photo review comparing the pre-treatment and post-treatment photographs. | 140 days (Arms A & B); 119 days (Arm C)
  Physician board-certified dermatologist to evaluate contour improvement per the Global Aesthetic Improvement Scale (GAIS), with scores in order of 'most improved' to 'worse': Most improved (score of 5); Much improved (score of 4); Improved (score of 3); No change (score of 2); Worse (score of 1).

SECONDARY OUTCOMES:
Blinded Investigator review comparing the pre-treatment photographs and post-treatment Follow-up live assessment. | Follow-up 1: 84 days (Arm A & B); 63 days (Arm C). Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Primary Investigator to evaluate live contour improvement compared to pre-treatment photographs per the Global Aesthetic Improvement Scale (GAIS), with scores in order of 'most improved' to 'worse': Most improved (score of 5); Much improved (score of 4); Improved (score of 3); No change (score of 2); Worse (score of 1).
Change in the subject Body Satisfaction Questionnaire (BSQ) | Follow-up 1: 84 days (Arm A & B); 63 days (Arm C). Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Subject self evaluation of the BSQ post treatment compared to Baseline with a possible score of: 5 (Very Satisfied); 4 (Satisfied); 3 (Neither Satisfied or Dissatisfied); 2 (Dissatisfied); and 1 (Very Dissatisfied).
Change in Anthropometric measurements: Abdominal Circumference | Treatment 1 and 3; Day 0 and Day 28 (Arm A and B). Treatment 1 and 5; Day 0 and Day 28 (Arm C). Follow-up 1: 84 days (Arm A & B); 63 days (Arm C). Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Pre- and post-treatment circumference (centimeters) changes made at Treatments 1 & 3 (Arm A & B) and Treatments 1 & 5 (Arm C). Follow-up visit circumference (centimeters) made at 1 and 3 months post treatment compared to baseline (All Arms).
Change in Anthropometric measurements: Abdominal Skinfold Thickness | Treatment 1; Day 0 (All Arms). Follow-up 1: 84 days (Arm A & B); 63 days (Arm C). Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Pre- and post-treatment abdominal skinfold thickness (millimeters) changes made at Treatment 1. Follow-up visit abdominal skinfold thickness (millimeters) changes made at one and three months post-treatment compared to baseline (All Arms).
Change in Anthropometric measurements: Weight | Treatment 1; Day 0 (All Arms). Follow-up 1: 84 days (Arm A & B); 63 days (Arm C). Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Pre- and post-treatment weight measurement (kg/lbs) changes made at Treatment 1. Follow-up visit weight measurement (kg/lbs) changes made at one and three months post-treatment compared to baseline (All Arms).

OTHER OUTCOMES:
Change in Abdominal Ultrasound images (optional) | Follow-up 1: 84 days (Arm A & B); 63 days (Arm C). Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Abdominal fat and muscle thickness (millimeters) changes from baseline to Follow-up 1 & 2 post last treatment as assessed using abdominal US images, compared to baseline.
Change in Abdominal Magnetic Resonance Imaging (MRI) (optional) | Follow-up 2: 140 days (Arms A & B); 119 days (Arm C)
  Abdominal fat and muscle thickness (millimeters) changes from baseline to Follow-up 2 post last treatment as assessed using MRI, compared to baseline.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scripps Clinical Research - General Medicine, San Diego, California
  - Schweiger Dermatology Group, Hackensack, New Jersey
  - Tennessee Clinical Research Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No